CLINICAL TRIAL: NCT01425853
Title: Non-Inferiority Clinical Trial On The Efficacy And Safety Of Chondroitin Sulfate And Glucosamine Hydrochloride In Combination Versus Celecoxib In Patients With Knee Osteoarthritis
Brief Title: Study on Efficacy and Safety of Chondroitin Sulfate + Glucosamine Hydrochloride Versus Celecoxib in Knee Osteoarthritis
Acronym: MOVES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRO/IV-ART-01; 2010-024010-61 (EudraCT Number)
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Chondroitin; Glucosamine; Chondroitin Sulfates; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chondroitin/Glucosamine (Droglican) (Experimental): Active ingredients: Chondroitin sulfate, 200 mg and Glucosamine hydrochloride 250 mg.
  Pharmacotherapeutic group: Other specific antirheumatic agents. Anatomical Therapeutic Chemical Classification System (ATC) code: M01CX.
  Interventions: Drug: Chondroitin/Glucosamine (Droglican)
- Celecoxib (Active Comparator): Active ingredient: Celecoxib, 200 mg. Pharmacotherapeutic group: Coxibs. ATC code: M01AH.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Chondroitin/Glucosamine (Droglican) — Experimental
  Other Names: Chondroitin sulfate/ Glucosamine hydrochloride
  Arms: Chondroitin/Glucosamine (Droglican)
Drug: Celecoxib — Active comparator
  Arms: Celecoxib

SUMMARY:
The purpose of this study is to determine whether the combination of Chondroitin sulfate (CS) and Glucosamine Hydrochloride (GH) has similar efficacy to Celecoxib (CE) in the treatment of patients with moderate to severe knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The primary objective of this study is to show that the combination treatment CS/GH has comparable efficacy to CE in pain reduction from baseline to 6 months of treatment measured with the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain subscale in knee OA patients with moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age
* Primary OA of the knee according to the American College of Rheumatology (ACR) criteria
* OA of radiological stages II or III according to Kellgren and Lawrence
* Patients with moderate-severe knee pain

Exclusion Criteria:

* Subjects with active malignancy of any type or history of a malignancy within the last five years
* Concurrent arthritic disease (antecedents and/or current signs) that could confound or interfere with the evaluation of pain efficacy such as chondrocalcinosis, Paget's disease of the ipsilateral limb to the target knee, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis seronegative spondylo-arthropathy, mixed connective tissue disease, collagen vascular disease, psoriasis, inflammatory bowel disease
* Pain in other parts of the body greater than the knee pain that could interfere with the evaluation of the index joint
* Patients with fibromyalgia
* Subjects with a history of heart attack or stroke, or who have experienced chest pain related to heart disease, or who have had serious diseases of the heart
* Subjects with high risk of cardiovascular (CV) events
* Subjects with any active acute or chronic infections requiring antimicrobial therapy, or serious viral (e.g., hepatitis, herpes zoster, HIV positivity) or fungal infections
* Subjects with a history of recurrent Upper Gastrointestinal (UGI) ulceration or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a significant coagulation defect
* Subjects who have been diagnosed as having or have been treated for oesophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to receiving the first dose of study medication
* Washout period for OA treatments before beginning the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Monfort, MD, Principal Investigator — Principal Investigator
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hochberg MC, Martel-Pelletier J, Monfort J, Moller I, Castillo JR, Arden N, Berenbaum F, Blanco FJ, Conaghan PG, Domenech G, Henrotin Y, Pap T, Richette P, Sawitzke A, du Souich P, Pelletier JP; MOVES Investigation Group. Combined chondroitin sulfate and glucosamine for painful knee osteoarthritis: a multicentre, randomised, double-blind, non-inferiority trial versus celecoxib. Ann Rheum Dis. 2016 Jan;75(1):37-44. doi: 10.1136/annrheumdis-2014-206792. Epub 2015 Jan 14. PMID 25589511

RESULTS

PARTICIPANT FLOW:
Groups:
- Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican): Active ingredients: Chondroitin sulfate, 200 mg and Glucosamine hydrochloride 250 mg.
  Pharmacotherapeutic group: Other specific antirheumatic agents. ATC code: M01CX.
  Chondroitin sulfate/ Glucosamine hydrochloride
- Celecoxib: Active ingredient: Celecoxib, 200 mg. Pharmacotherapeutic group: Coxibs. ATC code: M01AH.
  Celecoxib
Period: Overall Study
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Started | 304 | 302
Safety Population | 304 | 299
Per Protocol (PP) | 264 | 258
Completed | 240 | 225
Not Completed | 64 | 77

BASELINE CHARACTERISTICS:
Population: PP population was defined as all randomized patients who met the inclusion criteria, received study medication, had a baseline efficacy measurement and at least one corresponding post-baseline efficacy measurement (for the main efficacy variable) and did not present major violations of the protocol (n=522).
Groups:
- Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican): Active ingredients: Chondroitin sulfate, 200 mg and Glucosamine hydrochloride 250 mg.
  Pharmacotherapeutic group: Other specific antirheumatic agents. Anatomical Therapeutic Chemical Classification System (ATC) code: M01CX.
  Chondroitin sulfate/ Glucosamine hydrochloride
- Total: Total of all reporting groups
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib | Total
Number analyzed (Participants) | 264 | 258 | 522
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.22 (8.81) | 63.16 (9.02) | 62.68 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 209 | 438
  Male | 35 | 49 | 84
WOMAC Pain Subscale [Mean (Standard Deviation); unit: units on a scale] — Western Ontario & McMaster Universities Osteoarthritis Index, from 0 No Pain to 500 Maximum Pain
  units on a scale | 371.97 (41.76) | 370.60 (41.15) | 371.29 (41.57)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Pain Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale Score Range: 0 (no pain) - 500 (maximum pain) The study was designed such that the outcome of primary interest is knee pain related to OA. The measure selected to best evaluate this is an improvement in the WOMAC pain subscales. This subscale consists of 5 items which assesses the pain during walking, using stairs, in bed, sitting or lying, and standing.
Time Frame: 6 months
Population: Imputed data on PP population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale | 185.79 (7.43) | 184.67 (7.60)

2. Secondary Outcome: WOMAC Stiffness Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index, from 0 No Stiffness to 200 Maximum Stiffness WOMAC stiffness subscale was used to measure the stiffness of the knee with pain. Two items are used to assess stiffness grade: after first waking and later in the day.
Time Frame: 6 months
Population: ADO on PP population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale
  Baseline | 130.15 (34.97) | 129.48 (37.18)
  180 days | 69.06 (2.92) | 65.78 (2.99)

3. Secondary Outcome: WOMAC Function Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index, from 0 No Function to 1700 Maximum Function WOMAC functional limitation subscale was used to measure the functionality of the knee with pain. Seventeen items are used to assess functionality of the knee: tair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale
  Baseline | 1131.40 (242.68) | 1111.60 (267.81)
  180 days | 616.96 (23.51) | 595.78 (24.10)

4. Secondary Outcome: Huskisson's VAS
Description: Visual Analogue Scale: 0 No Pain 100 Maximum Pain Huskisson's VAS measures global pain intensity. Patients were asked to quantify their disease status on a 100 mm VAS as follows: "Please indicate the severity of knee pain experienced during the last 48 hours by marking a (I) through the line". Left hand marker represents "No pain" and right hand marker represents "The worst pain imaginable".
Time Frame: 6 months
Population: ADO on PP population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale
  Baseline | 72.79 (15.12) | 73.47 (15.10)
  180 days | 37.86 (1.61) | 37.64 (1.65)

5. Secondary Outcome: Percentage of Participants With Response as Defined by Outcome Variables for Osteoarthritis Clinical Trials - Osteoarthritis Research Society International (OMERACT-OARSI)
Description: The OARSI Standing Committee for Clinical Trials Response Criteria Initiative and the OMERACT committee, in concert with the international rheumatology community, has led to the development of a uniform core set of outcome measures for OA. One of the objectives was to propose a set of criteria for measurement based on multiple domains to present the results of changes after treatment in symptomatic parameters as a single variable for clinical trials.
  To be considered as responder patients should met one the following criteria:
  * High improvement in pain or in function ≥ 50% and absolute change ≥ 20 or
  * Improvement in at least 2 of the 3 following:
    * Pain ≥ 20% and absolute change ≥ 10
    * Function ≥ 20% and absolute change ≥ 10
    * Patient's global assessment ≥ 20% and absolute change ≥ 10
Time Frame: 6 months
Population: ADO on PP population
Measure: Number; unit: percentage of participants
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 236 | 221
percentage of participants | 79.7 | 79.2

6. Secondary Outcome: Percentage of Presence of Joint Swelling
Description: Study knees were evaluated at each visit for the presence or absence of swelling and/or effusion.
Time Frame: 6 months
Population: ADO on PP population
Measure: Number; unit: percentage of participants
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 236 | 221
percentage of participants | 5.9 | 4.5

7. Secondary Outcome: Percentage of Presence of Joint Effusion
Description: Study knees were evaluated at each visit for the presence or absence of swelling and/or effusion.
Time Frame: 6 months
Population: ADO on PP population
Measure: Number; unit: percentage of participants
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 236 | 221
percentage of participants | 4.1 | 3.8

8. Secondary Outcome: Consumption of Rescue Medication
Description: Use of rescue medication as number of paracetamol tablets 500 mg since the last visit. The tablet count was reconciled with the patient diary.
  Total Number of pills per month
Time Frame: 6 months
Population: Consumption of rescue medication (number of daily tablets consumed). ADO on PP population. daily tablets consumed/month
Measure: Mean (Standard Deviation); unit: daily tablets consumed/month
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
daily tablets consumed/month | 31.0 (2.6) | 29.0 (2.7)

9. Secondary Outcome: Patient's Global Assessment (PGA) and Investigator's Global Assessment (IGA) of Disease Activity
Description: Patients were asked to quantify their disease status on a VAS scale with range 0 mm (best) and 100 mm (worst) as follows: "Considering all the ways your arthritis of the knee affects you, mark (I) on the scale how well you are doing." Left hand marker "Very Well", Right hand marked "Very Poor".
Time Frame: 6 months
Population: Patient and Investigator's global assessment of disease activity. ADO on PP population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale
  PGA Activity Baseline | 69.11 (17.34) | 69.41 (16.44)
  PGA Activity 180 days | 38.35 (1.54) | 36.88 (1.59)
  IGA Activity Baseline | 63.2 (15.54) | 63.28 (14.71)
  IGA Activity 180 daus | 35.33 (1.39) | 33.40 (1.42)

10. Secondary Outcome: Patient's and Investigator's Global Assessment of Response to Therapy
Description: The investigator were asked to evaluated the patient's response to therapy of the index knee by marking a (I) a VAS scale with range 0 mm (best) and 100 mm (worst) as follows: Left hand marker "Excellent-Best possible anticipated response, considering the severity and stage of the disease", right hand marker "None-no response, absence of drug effect".
Time Frame: 6 months
Population: Investigator and Patient's global assessment assessment of response to therapy. ADO on PP population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
units on a scale
  PGA Therapy Baseline | 54.59 (1.55) | 45.9 (1.57)
  PGA Therapy 180 days | 36.85 (1.70) | 36.04 (1.75)
  IGA Therapy Baseline | 51.4 (1.43) | 42.25 (1.45)
  IGA Therapy 180 days | 34.72 (1.6) | 33.83 (1.64)

11. Secondary Outcome: Health Status According to EuroQoL
Description: EuroQoL-5D was a standardized instrument for use as a measure of health outcome that provides a simple descriptive profile and a single index value for health status. It was assessed at all of the study visits.
  The EQ-5D-3L essentially consists of 2 pages - the EQ-5D descriptive system (page 2) and the EQ visual analogue scale (EQ VAS) (page 3). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. Total scale range for each dimension reported is 1 to 3.
  The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
  Total scale range for VAS dimension reported is 0 to 100.
Time Frame: 6 months
Population: ADO on PP population
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 264 | 258
points
  Mobility Baseline | 1.84 (0.37) | 1.84 (0.38)
  Mobility 180 Days | 1.52 (0.033) | 1.46 (0.034)
  Self-care Baseline | 1.39 (0.49) | 1.44 (0.5)
  Self-care 180 days | 1.19 (0.026) | 1.21 (0.027)
  Usual activities Baseline | 1.78 (0.44) | 1.79 (0.42)
  Usual activities 180 days | 1.42 (0.033) | 1.42 (0.034)
  Pain Discomfort Baseline | 2.25 (0.43) | 2.27 (0.45)
  Pain Discomfort 180 days | 1.84 (0.032) | 1.86 (0.033)
  Anxiety depression baseline | 1.70 (0.58) | 1.60 (0.58)
  Anxiety depression 180 days | 1.43 (0.038) | 1.34 (0.035)
  VAS Baseline | 54.545 (20.33) | 52.488 (20.66)
  VAS 180 days | 69.080 (1.28) | 70.219 (1.31)

12. Secondary Outcome: Number of Participants With at Least One Adverse Events
Description: The safety evaluation was done in the set of randomized patients who took at least one dose of the medication
Time Frame: 6 months
Population: Safety population
Measure: Number; unit: number of participants
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 304 | 299
number of participants | 155 | 151

13. Secondary Outcome: Number of Adverse Events Defined by Relationship With Treatment
Description: The safety evaluation was done in the set of randomized patients who took at least one dose of the medication
Time Frame: 6 months
Population: Safety population
Measure: Number; unit: number of events
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Number analyzed (Participants) | 304 | 299
number of events
  Treatment-related AEs: Definitive | 3 | 10
  Treatment-related AEs: Possibly | 43 | 38
  Treatment-related AEs: Probably | 25 | 12
  Treatment-related AEs: Non-appraisable | 0 | 1
  Treatment-related AEs: unlikely or unrelated | 84 | 90

14. Secondary Outcome: Biomarker Analysis
Description: The following biomarkers will be evaluated: COMP, Coll2-1, Coll2-1 NO2 and Fib3-2
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) | Celecoxib
Serious Adverse Events (participants affected / at risk) | 7/304 | 10/299
Other Adverse Events (participants affected / at risk) | 119/304 | 112/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) (N=304) | Celecoxib (N=299)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Obesity surgery (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chondroitin Sulfate/ Glucosamine Hydrochloride (Droglican) (N=304) | Celecoxib (N=299)
Abdominal Pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Tootache (Gastrointestinal disorders) | 3 (3) | 4 (4)
Bronchitis (Infections and infestations) | 10 (10) | 7 (7)
Cystitis (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 26 (30) | 23 (26)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 20 (27) | 9 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7)
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (3)
Headache (Nervous system disorders) | 25 (56) | 31 (93)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No